CLINICAL TRIAL: NCT00932191
Title: Endothelial Cell Loss After Cataract Surgery: Comparison of a Reduced Ultrasound Technique Versus Standard Ultrasound Technique
Brief Title: Endothelial Cell Loss After Cataract Surgery
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Stopped for lack of funds
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DHCrush001
Record Dates: First submitted 2009-07-01; First posted 2009-07-03 (Estimated); Last update posted 2014-08-25 (Estimated); Status verified 2014-08

CONDITIONS: Cataracts
Keywords: Cataract; Corneal endothelial cell loss; Ultrasound power; Corneal endothelium
MeSH Terms: conditions — Cataract; Corneal Endothelial Cell Loss

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ultrasound phacoemulsification (Active Comparator): Cataract nucleus is removed using standard amounts of ultrasound energy.
  Interventions: Procedure: Standard phacoemulsification
- Reduced ultrasound phacoemulsification (Active Comparator): Cataract nucleus removal using less ultrasound energy and more mechanical energy.
  Interventions: Procedure: Reduced ultrasound phacoemulsification

INTERVENTIONS:
Procedure: Standard phacoemulsification — Cataract nucleus removal using standard amounts of ultrasound energy
  Arms: Ultrasound phacoemulsification
Procedure: Reduced ultrasound phacoemulsification — Cataract nucleus removal using less ultrasound energy and more mechanical energy.
  Arms: Reduced ultrasound phacoemulsification

SUMMARY:
The purpose of this study is to compare two cataract surgical technique variations for removing the nucleus of the lens (central part of the lens) in terms of damage to the inner layer of the cornea which is called the endothelium. One variation uses more ultrasound energy and the other more mechanical force to break up the nucleus.

ELIGIBILITY:
Inclusion Criteria:

* Visually significant moderate density cataract

Exclusion Criteria:

* Corneal or retinal pathology limiting visual potential to worse than 20/40
* Lens pathology including pseudoexfoliation or lens dislocation
* Prior intraocular surgery
* Age less than 40

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2009-07; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Corneal endothelial cell loss by specular microscopy after cataract surgery | 3 months post-operatively

CONTACTS AND LOCATIONS:
Overall Officials: David Hwang, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States